CLINICAL TRIAL: NCT07397286
Title: Comparison of the Efficacy of Combined Dorsal Root Ganglion Pulsed Radiofrequency and Cervical Transforaminal Epidural Steroid Injection With and Without Local Anesthetic in Cervical Disc Herniation, Prospective Controlled Study
Brief Title: The Effect of Adding a Local Anesthetic to Transforaminal Epidural Injection in Cervical Disc Herniation.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Esra Ertilav, Assoc. Prof., Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025/297
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Transforaminal Epidural Injection; Dorsal Root Ganglion Stimulation; Servical Disc Herniation
MeSH Terms: interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients to whom applied epidural injection with local anaesthetic (Experimental): Patients in Group 1 are given 4 mg of dexamethasone + 20 mg of lidocaine. The radiofrequency generator is adjusted so that the catheter needle tip temperature does not exceed 42 ºC, and they undergo pulsed radiofrequency treatment for 4 minutes
  Interventions: Procedure: servical transforaminal epidural steroid injection with local anaesthetic
- patients to whom applied epidural injection without local anaesthetic (Active Comparator): Patients in Group 2 are given 4 mg of dexamethasone. The radiofrequency generator is adjusted so that the catheter needle tip temperature does not exceed 42 ºC, and they undergo pulsed radiofrequency treatment for 4 minutes.
  Interventions: Procedure: servical transforaminal epidural steroid injection without local anaesthetic

INTERVENTIONS:
Procedure: servical transforaminal epidural steroid injection with local anaesthetic — The interventional treatment procedure is performed in the operating room under sterile conditions, in the supine position, using a C-arm fluoroscopy device.Subsequently, patients in Group 1 receive 4 mg dexamethasone and 1cc lidocain. The radiofrequency generator is adjusted so that the temperature of the catheter needle tip does not exceed 42 ºC.
  Arms: patients to whom applied epidural injection with local anaesthetic
Procedure: servical transforaminal epidural steroid injection without local anaesthetic — The interventional treatment procedure is performed in the operating room under sterile conditions, in the supine position, using a C-arm fluoroscopy device.Subsequently, patients in Group 2 receive 4 mg dexamethasone. The radiofrequency generator is adjusted so that the temperature of the catheter needle tip does not exceed 42 ºC.
  Arms: patients to whom applied epidural injection without local anaesthetic

SUMMARY:
The study is designed as a double-blind, prospective, randomized controlled trial. Blindness is ensured by having different researchers performing the interventional procedures and monitoring the pain diaries, thus preventing them from knowing which procedure is performed on which patient. Patient randomization will be performed using computer assistance.

After obtaining approval from the hospital ethics committee, clinical trials will be initiated. Patients who present to the Department of Neurology, Algology Division, ADÜTF between 2025-2026 and undergo DRG-PRF and TFAESI for radicular pain due to cervical disc herniation will be divided into two groups. Patients in Group 1 will undergo DRG-PRF and TFAESI with the addition of local anesthetic. Patients in Group 2 will undergo DRG-PRF and TFAESI without the addition of local anesthetic. During the study, NRS score measurements will be taken to assess pain intensity in patients in both Group 1 and Group 2 before the procedure and at 1, 3, and 6 months post-procedure follow-ups. Neurological and musculoskeletal examinations will be performed during routine check-ups before the procedure and at 1, 3, and 6 months after the procedure, and any developing side effects will be recorded.

DETAILED DESCRIPTION:
The interventional treatment procedure is performed in the operating room under sterile conditions, in the supine position, using a C-arm fluoroscopy device. The first intervertebral foramen visible under fluoroscopy is C2-C3. Once the appropriate cervical space is identified, the C-arm fluoroscopy device is directed obliquely to 45-65 degrees until the cervical neural foramen is visualized as a circle. The cannula insertion site is determined. The skin and subcutaneous tissue are anesthetized with 2% lidocaine. A 5 cm long RF cannula with a 5 mm active tip is advanced towards the 6 o'clock position of the neural foramina. The needle is advanced until it contacts the superior facet joint, then guided into the foramen. After entering the foramen, to avoid direct intrathecal or spinal cord damage, the needle is advanced to the facet column and into the epidural space while anteroposterior views are obtained with fluoroscopy. Approximately 0.5 mL of non-ionizing contrast agent is injected to confirm needle placement. The spread of radiopaque material, which adheres to the periradicular membrane, is observed both within the foramen and around the nerve root during fluoroscopy. If abnormal sensation, vibration, or pain is observed with a stimulus less than 0.7 Volts for sensory stimulation, or if a pulse is felt in the arm with a stimulus less than 2.0 Volts for motor stimulation, it is assumed that the catheter needle has been placed near the dorsal root ganglion. Subsequently, patients in Group 1 are given 4 mg dexamethasone + 20 mg lidocaine, and patients in Group 2 are given 4 mg dexamethasone. The radiofrequency generator is adjusted so that the temperature of the catheter needle tip does not exceed 42 ºC, and it is subjected to pulsed radiofrequency treatment for 4 minutes. Patient response will be determined based on the reduction in pain at follow-up examinations at 1, 3, and 6 months after the procedure as follows: good response > 50% reduction, poor response < 50% reduction, or no change, no response.

ELIGIBILITY:
Inclusion Criteria:

* Patients consisted of those who presented to our outpatient clinic with neck and arm pain, who had received medical and/or physical therapy but whose symptoms did not improve.

Exclusion Criteria:

* The procedure was not performed on those with neurological deficits requiring surgery, those with known allergies to lidocaine and dexamethasone, those who had recently undergone head and neck surgery, diabetic patients with impaired blood sugar regulation, those who had received epidural steroid injections or depot steroids within the last 15 days, those with progressive neurological deficits, those with coagulation disorders (INR > 1.5; platelets < 100,000/mm³), those with any lesion or infection in the cervical region that would prevent epidural intervention, and pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
To compare whether the addition of a local anesthetic to combined DRG-pulsed RF and transforaminal anterior epidural steroid injection (TAESI) treatment makes a difference in clinical efficacy in patients with cervical disc herniation | 6 months
  In patients with radicular neck pain due to cervical disc herniation, the clinical efficacy of adding a local anesthetic during combined DRG-pulsed RF and transforaminal anterior epidural steroid injection (TAESI) was evaluated using the NRS (Numerical Rating Scale) to assess pain control.

CONTACTS AND LOCATIONS:
Locations (1):
- Adnan Menderes University Efeler / Aydın, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No